CLINICAL TRIAL: NCT04907097
Title: Effect of Monomeric and Oligomeric Flavanols on Exercise Blood Pressure and Vascular Function in Healthy Volunteers
Brief Title: Effect of MOF on Exercise Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: VieCuri Medical Centre (Other); CEP Group Holding B.V. (Unknown); Campus Venlo (Unknown)
Responsible Party: Principal Investigator, Khrystyna Semen, Professor assistant, Maastricht University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: NL77344.068.21
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: Vascular function; Monomeric and oligomeric flavanols; Grape seeds extract; Exercise blood pressure; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOF/placebo (Other): During period 1 (4 weeks) participants will receive monomeric and oligomeric flavanols and during period 2 (4 weeks) placebo. Wash out period between two interventions will be 4 weeks. The daily dose of monomeric and oligomeric flavanols will be 200 mg (2 capsules once a day) and for placebo (2 capsules once a day).
  Interventions: Dietary Supplement: Monomeric and oligomeric flavanols; Other: Placebo
- Placebo/MOF (Other): During period 1 (4 weeks) participants will receive placebo and during period 2 (4 weeks) monomeric and oligomeric flavanols. The wash out period between two interventions will be 4 weeks. The daily dose of placebo will be 2 capsules once a day and for monomeric and oligomeric flavanols 200 mg (2 capsules once a day).
  Interventions: Dietary Supplement: Monomeric and oligomeric flavanols; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Monomeric and oligomeric flavanols — Monomeric and oligomeric flavanols will be derived from Vitis vinifera seeds extract.
  Other Names: Masquelier's original OPCs
Other: Placebo — Placebo capsuled will be used as a comparator.

SUMMARY:
The purpose of this study is to establish an effect of monomeric and oligomeric flavanols supplementation on exercise blood pressure and vascular function in healthy volunteers.

DETAILED DESCRIPTION:
Exaggerated exercise blood pressure (BP) response in healthy subjects is recognized as a risk factor of hypertension and cardiovascular events. Pathogenetically exaggerated BP response is attributed to compromised vascular(endothelial) functions as well as oxidative stress and inflammation. Monomeric and oligomeric flavanols (MOF) are dietary components with well-characterized beneficial effects on the redox homeostasis, endothelial function and microvascular health.

The objectives of the study will be to evaluate the effects of MOF in comparison to placebo on exercise blood pressure, endothelial function, inflammatory and redox status in healthy prehypertensive volunteers. In addition, the study will aim to assess the impact of MOF supplementation on the exercise-induced renin-angiotensin-aldosterone system (RAAS) activation and extracellular matrix remodelling.

After being informed about the study and potential risks all volunteers signing informed consent form will undergo screening to determine eligibility for the study. Eligible subjects will be randomized in the double-blind manner to monomeric and oligomeric flavanols /placebo or placebo/monomeric and oligomeric flavanols sequence (cross-over design) in a 1:1 ratio. Monomeric and oligomeric flavanols are derived from grape seeds extract and will be administered in a dose 200 mg per day.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women with normal to high-normal resting BP (SBP 120 - 139 mm Hg and DBP 80 - 89 mm Hg).
2. Age 35 - 65 years
3. BMI 20 - 32 kg/m^2
4. Hypertensive response to maximal exercise test defined as SBP ≥ 200 mm Hg (men) and ≥ 180 mm Hg (women).

Exclusion Criteria:

1. Active engagement in the weight loss programs, also including slimming diets.
2. Active smoking or abstinence from smoking for less than one year.
3. Use of medications that reduce BP and/or can potentially influence other study outcomes (ACE-inhibitors, angiotensin receptor blockers, diuretics, painkillers, etc).
4. Intake of polyphenol-containing supplements for two month before and during the whole course of the study.
5. History of diabetes, cardiovascular, respiratory, renal, gastrointestinal, hepatic or other diseases and conditions, which potentially can compromise participation in this study.
6. Intense sporting (>10 h/week) and/or participation in the competition at the professional level.
7. Pregnancy or breastfeeding.
8. Participation in a clinical trial within 4 weeks prior to inclusion into this study.
9. Vaccination against Covid-19 within two months before the screening/randomization visit or expected vaccination against Covid-19 during the study

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure from before to peak value during the submaximal exercise test | Day 28±3, Day 84±3
  Excessive increase in systolic blood pressure during exercise is a well-characterized risk-factor of cardiovascular disease and is related to signs of sub clinical endothelial dysfunction.
Change in mean blood pressure from before to peak value during the submaximal exercise test | Day 28±3, Day 84±3
  Increase in mean blood pressure during exercise is related to signs of endothelial dysfunction.

SECONDARY OUTCOMES:
Carotid-femoral pulse wave velocity | Day 28±3, Day 84±3
  Carotid-femoral pulse wave velocity reflects arterial stiffness and is related to the cardiovascular risk.
Biomarkers of RAAS activation | Day 28±3, Day 84±3
  Renin, angiotensin II and aldosterone are involved in regulation of blood pressure response also during exercise.
Biomarkers of inflammation | Day 28±3, Day 84±3
  High-sensitivity C-reactive protein (hs-CRP), interleukin (IL)-6, tumor necrosis factor-alpha (TNFalpha) are well-recognized molecules that characterize inflammation.
Biomarkers of oxidative stress | Day 28±3, Day 84±3
  Malondialdehyde (MDA), trolox equivalent antioxidant capacity (TEAC) reflect the activity lipid peroxidation and antioxidant defense and therefore are indicative about the condition of redox homeostasis.
Biomarkers of endothelial function | Day 28±3, Day 84±3
  Endothelin 1 and levels of nitrate/nitrite are commonly used to assess endothelial function and characterize balance between vasodilation and vasoconstriction.
Biomarkers of vascular remodelling | Day 28±3, Day 84±3
  Metalloproteinase (MMP)-9, MMP-2, tissue inhibitor of metalloproteinase (TIMP)-1, TIMP-4 are involved in modulation of extracellular matrix and their activity have been linked to vascular health.
Other hemodynamic parameters | Day 28±3, Day 84±3
  Values of systolic and diastolic blood pressure and heart rate at rest and during exercise recovery are indicators of cardiovascular risk and were related also to hemodynamic response during peak exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Khrystyna O. Semen, MD, PhD, Principal Investigator — Professor assistant
Locations (1):
- VieCuri Medical Center, Venlo, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No